CLINICAL TRIAL: NCT00861692
Title: An Open-label, Multi-centre, Clinical Study to Collect Information on the Clinical Use of Argatroban in Patients With Heparin Induced Thrombocytopenia (HIT) Type II Who Require Parenteral Antithrombotic Therapy
Brief Title: Clinical Management of Argatroban in Patients With Heparin Induced Thrombocytopenia Type II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARG-E07
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Heparin-induced Thrombocytopenia Type II
Keywords: Argatroban; heparin induced thrombocytopenia (HIT); direct thrombin inhibitor (DTI)
MeSH Terms: interventions — argatroban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Argatroban (Experimental)
  Interventions: Drug: argatroban

INTERVENTIONS:
Drug: argatroban

SUMMARY:
The purpose of this study is to collect data on the clinical management of Argatroban in patients with suspected or confirmed heparin-induced thrombocytopenia Type II, with or without ongoing thrombosis who require parenteral antithrombotic therapy

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged >= 18 years
* Females of child bearing potential must have a negative urine pregnancy test prior to entry into the study
* Patients with suspected or confirmed heparin-induced thrombocytopenia Type II, with or without ongoing thrombosis who require parenteral anticoagulation
* Signed written informed consent by the subject, or if the subject is unable to do so, consent will be sought from their family member, or a trusted person nominated by the subject or the legal representative

Exclusion Criteria:

* Uncontrolled bleeding
* Severe hepatic impairment (Child-Pugh Class C)
* Hypersensitivity to argatroban or to any of the excipients (sorbitol and ethanol)
* Pregnancy (exclusion by routine urine test)
* Lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Principal Investigator — Information at Mitsubishi Pharma Europe
Locations (1):
- Saint-Etienne, France

REFERENCES:
- [Result] Tardy-Poncet B, Nguyen P, Thiranos JC, Morange PE, Biron-Andreani C, Gruel Y, Morel J, Wynckel A, Grunebaum L, Villacorta-Torres J, Grosjean S, de Maistre E. Argatroban in the management of heparin-induced thrombocytopenia: a multicenter clinical trial. Crit Care. 2015 Nov 11;19:396. doi: 10.1186/s13054-015-1109-0. PMID 26556106

RESULTS

PARTICIPANT FLOW:
Groups:
- Argatroban: start with 1μg/kg/min infusion to be adjusted to aPTT 1.5-3.0 times the baseline values
Period: Overall Study
Arm/Group | Argatroban
Started | 20
Completed | 14
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | Argatroban
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Composite of All-cause Death, Thrombosis (New and Extended) and Unplanned Amputation
Time Frame: During and 30 days after argatroban treatment
Measure: Number; unit: participants
Arm/Group | Argatroban
Number analyzed (Participants) | 20
participants | 10

2. Primary Outcome: All-cause Death
Time Frame: During and 30 days after argatroban treatment
Measure: Number; unit: participants
Arm/Group | Argatroban
Number analyzed (Participants) | 20
participants | 6

3. Primary Outcome: Death Related to Heparin-induced Thrombocytopenia (HIT)
Time Frame: During and 30 days after argatroban treatment
Measure: Number; unit: participants
Arm/Group | Argatroban
Number analyzed (Participants) | 20
participants | 0

4. Primary Outcome: Number of Patients With Thrombosis (New and Extended)
Time Frame: During and 30 days after argatroban treatment
Measure: Number; unit: participants
Arm/Group | Argatroban
Number analyzed (Participants) | 20
participants | 5

5. Primary Outcome: Number of Patients With Unplanned Amputation
Time Frame: During and 30 days after argatroban treatment
Measure: Number; unit: participants
Arm/Group | Argatroban
Number analyzed (Participants) | 20
participants | 0

6. Primary Outcome: Number of Patients With Major or Minor Bleeding
Description: Major bleeding is defined as i) overt and associated with a fall in the haemoglobin level 2 g/dl or more, ii) leads to transfusion of 2 units or more, iii) is retroperitoneal, iv) occurs into a major prosthetic joint, or v) in intracranial.
  Minor bleeding is defined as overt bleeding that does not meet the criteria of major bleeding.
Time Frame: During and 30 days after argatroban treatment
Measure: Number; unit: participants
Arm/Group | Argatroban
Number analyzed (Participants) | 20
participants | 4

7. Primary Outcome: Number of Patients With Platelet Count Recovery
Description: Platelet increase of ≥ 100G/L or 50%.
Time Frame: Day 3
Population: Data are missing in 3 patients.
Measure: Number; unit: participants
Arm/Group | Argatroban
Number analyzed (Participants) | 17
participants | 12

ADVERSE EVENTS:
Arm/Group | Argatroban
Serious Adverse Events (participants affected / at risk) | 14/20
Other Adverse Events (participants affected / at risk) | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Argatroban (N=20)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1
CARDIAC ARREST (Cardiac disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1
MYOCARDIAL RUPTURE (Cardiac disorders) | 1
PERITONITIS (Gastrointestinal disorders) | 2
COLITIS (Gastrointestinal disorders) | 1
HAEMATEMESIS (Gastrointestinal disorders) | 1
PNEUMATOSIS INTESTINALIS (Gastrointestinal disorders) | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1
MULTI-ORGAN FAILURE (General disorders) | 1
SEPSIS (Infections and infestations) | 3
SEPTIC SHOCK (Infections and infestations) | 1
MEDICATION ERROR (Injury, poisoning and procedural complications) | 1
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1
BLUE TOE SYNDROME (Vascular disorders) | 1
FEMORAL ARTERY EMBOLISM (Vascular disorders) | 1
HAEMORRHAGE (Vascular disorders) | 1
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Argatroban (N=20)
Anaemia (Blood and lymphatic system disorders) | 7
Coagulopathy (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 3
Bradycardia (Cardiac disorders) | 2
Mitral Valve Incompetence (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Colonic Polyp (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Impaired Gastric Emptying (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Rectal Haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Chest Pain (General disorders) | 1
Generalised Oedema (General disorders) | 1
Hyperthermia (General disorders) | 2
Inflammation (General disorders) | 2
Injection Site Inflammation (General disorders) | 1
Malaise (General disorders) | 1
Oedema Peripheral (General disorders) | 2
Pain (General disorders) | 4
Puncture Site Haemorrhage (General disorders) | 1
Pyrexia (General disorders) | 4
Cholestasis (Hepatobiliary disorders) | 2
Hepatic Function Abnormal (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Jaundice Cholestatic (Hepatobiliary disorders) | 1
Liver Disorder (Hepatobiliary disorders) | 1
Hypogammaglobulinaemia (Immune system disorders) | 1
Device Related Infection (Infections and infestations) | 4
Escherichia Urinary Tract Infection (Infections and infestations) | 2
Fungal Infection (Infections and infestations) | 1
Fungal Sepsis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Postoperative Wound Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Haemodialysis Complication (Injury, poisoning and procedural complications) | 1
Incision Site Pain (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 3
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1
Alpha Globulin Increased (Investigations) | 1
Blood Pressure Decreased (Investigations) | 1
Coagulation Time Prolonged (Investigations) | 2
Cytomegalovirus Test Positive (Investigations) | 1
Globulins Decreased (Investigations) | 1
Glomerular Filtration Rate Increased (Investigations) | 1
Haemoglobin Decreased (Investigations) | 2
International Normalised Ratio Increased (Investigations) | 2
Pulmonary Function Test Decreased (Investigations) | 2
Transaminases Increased (Investigations) | 1
Weight Decreased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Folate Deficiency (Metabolism and nutrition disorders) | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Hypovolaemia (Metabolism and nutrition disorders) | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2
Altered State Of Consciousness (Nervous system disorders) | 1
Depressed Level Of Consciousness (Nervous system disorders) | 1
Monoparesis (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional State (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Sleep Disorder (Psychiatric disorders) | 1
Calculus Bladder (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Renal Impairment (Renal and urinary disorders) | 1
Acute Lung Injury (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 1
Skin Dystrophy (Skin and subcutaneous tissue disorders) | 1
Aortic Arteriosclerosis (Vascular disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Haemodynamic Instability (Vascular disorders) | 3
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 5
Venous Thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other